CLINICAL TRIAL: NCT03564522
Title: Image-based Multi-scale Modeling Framework of the Cardiopulmonary System: Longitudinal Calibration and Assessment of Therapies in Pediatric Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Michigan State University (Other); Nationwide Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alberto Figueroa, Edward B Diethrich M.D. Research Professor of Biomedical Engineering and Vascular Surgery, University of Michigan
Other Study IDs: HUM00117706; U01HL135842 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-06-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension; Congenital Heart Disease; Pediatric Congenital Heart Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Defects, Congenital | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Hypertension: Participants diagnosed with pulmonary hypertension that will undergo a clinically indicated cardiac catheterization and cMRI.
  Interventions: Procedure: cardiac catheterization; Radiation: Cardiac MRI
- Heart Transplant: Successful cardiac transplant recipient without evidence of pulmonary hypertension, that will undergo clinically indicated cardiac catheterization.
  Interventions: Procedure: cardiac catheterization; Radiation: Cardiac MRI

INTERVENTIONS:
Procedure: cardiac catheterization — cardiac catheterizations will be clinically indicated and the study will collect this clinical data.
Radiation: Cardiac MRI — If clinically indicated, the study will collect data from MRIs.

SUMMARY:
This study looks to develop a multi-scale computational model of Pulmonary Hypertension, this clinical model will be calibrated using longitudinal, retrospectively and prospectively acquired human clinical data.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a complex disorder associated with elevated pulmonary arterial pressure. Unlike systemic hypertension, PH is difficult to detect in routine physical examinations and the current gold standard for diagnosing PH is through invasive right heart catheterization. Prolonged PH results in functional, structural and anatomical changes in the right ventricle (RV), large pulmonary arteries, and the pulmonary micro-circulation that ultimately lead to decompensated RV failure and death. Unlike in systemic hypertension, for which patients have effective pharmacological management of blood pressure for decades, PH prognosis remains poor with 15% mortality within 1 year on modern therapy. Our current understanding of PH has largely been obtained through animal models and clinical studies. However, surgical banding or chronic hypoxia animal models do not fully reproduce the etiology of human PH, whereas invasive clinical measurements of pulmonary vascular resistance (PVR), stiffness and ventricular elastance provide limited insight into disease progression. Therefore, there is a pressing need to develop a multi-scale (MS) computational model that can couple the short term (e.g. hemodynamics) and long-term G&R interactions between the RV and the pulmonary circulation.

The overall goals of this project are to use the framework to (1) describe the time course of the biomechanical alterations and (2) identify the key mechanical culprits associated with PH-induced heart failure so that clinical interventions can be targeted against them.

ELIGIBILITY:
Inclusion Criteria:

* Patients has been clinically diagnosed with pulmonary hypertension (>25 mmHg) or patient is a biopsy-proven non-rejecting cardiac transplant recipient
* Receiving partial or full care from pediatric cardiology team at Mott Children's Hospital (may have a primary cardiologist elsewhere).

Exclusion Criteria:

* Girls and women who are pregnant or actively trying to become pregnant
* Patients with significant neurocognitive impairment that precludes their ability to sign a consent form
* Patient has a contraindication to right-heart catheterization (RHC) examination, which includes patients with hypoxia and those who have difficulty maintaining supine position for the procedure.
* Patients with the following genetic syndromes:Trisomy 21 if unable to assent or consent, Trisomy 18,Trisomy 13, Other genetic syndromes at the discretion of the Primary Investigator
* Patients with unrepaired single ventricles (i.e., Pre-Fontan physiology)
* Patients who have heart failure and are deemed to be high risk to undergo tests that require sedation/anesthesia.
* Patients who require IV sedation or general anesthesia for research only MRI
* Patients with a pacemaker/internal defibrillator will be excluded from MRI PORTION ONLY

Ages: 6 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pulmonary hypertension patients will be defined by a mean artery blood pressure >25 mmHg. Transplant patients are tested for pulmonary vascular resistance prior to transplant; if it is too high, transplant is contraindicated. So this group comprises patients who have normal right ventricular function and pulmonary vascular function to act as a control for the right-sided disease that we are testing, and in addition regularly undergo cardiac catheterization for clinical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
3D volumetric data (mL/m2) | 1 hour
  Modeling framework will be validated using 3D volumetric data (mL/m2) gathered via cardiac MRI
Cardiopulmonary Flow (mL/beat) | 1 hour
  Modeling framework will be validated using cardiopulmonary flow (mL/beat) gathered via cardiac MRI
Mean Pressure (mmHg) | 2 hours
  Modeling framework will be validated using pressures (mmHg) gathered via cardiac catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Figueroa, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Mott Children's Hospital University of Michigan, Ann Arbor, Michigan
  - Nationwide Children's Hospital, Columbus, Ohio